



## Enhancing CAMHS Referrals 2 (EN-CAMHS 2) CONSENT FORM

Name of Researchers: Prof Kathryn Abel & Charlotte Stockton-Powdrell

If you are happy to participate, please complete and sign the consent form below

| No. | Activities | Initials |
|---|---|---|
| 1 | I confirm that I have read and understand the information sheet V2.1 30/10/2025 for the above study. I have had the opportunity to consider the information, ask questions, and have had these answered satisfactorily. | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason and without detriment to myself. I understand that if I withdraw, any data that has already been anonymised from my interview participation will still be used in the study. | |
| | I agree to take part on this basis. | |
| 3 | I agree to take part in the research activity to use the digital CAMHS referral tool. | |
| 4 | I agree for the research activity to be audio and video recorded and understand that the recording will be written out in full (transcribed) and any identifiable information will be removed. The audio and video recording will then be destroyed. | |
| 5 | I agree that any data collected may be included in anonymous form in publications/conference presentations (e.g., academic conferences, journals). I understand that this could include a direct quote from the research activity which has been anonymised (i.e. all identifiable information removed). | |
| 6 | I understand that data collected during the study may be looked at by responsible individuals from the University of Manchester, Greater Manchester Mental Health NHS Foundation Trust or regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to this data. | |
| 7 | I understand that this consent form and anonymised research data collected about me during this study will be retained for a period of five years after which it will be destroyed. | |
| 8 | I agree to take part in this research | |

V 2.1 30/10/2025 IRAS 332029





## **Optional:**

| 9 | I agree that the researchers may retain my contact | Yes / No |
|---|---|---|
| | details in order to provide me with a summary of the | |
| | findings for this study. | (delete as appropriate) |

**Data Protection** 

The personal information we collect and use to conduct this research will be processed in accordance with UK data protection law as explained in the Participant Information Sheet and the University of Manchester Privacy Notice for Research Participants.

| Please sign below: |
|------------------------------------|
| Name of participant: |
| Date: |
| Signature: |
| Name of the person taking consent: |
| Date: |
| Signature: |

V 2.1 30/10/2025 IRAS 332029